CLINICAL TRIAL: NCT00870519
Title: Evaluation of [123I] MNI-168 and SPECT as a Marker of Beta-amyloid Protein Deposition in Subjects With Alzheimer Disease in Comparison to Healthy Subjects
Brief Title: Brain Imaging Study in Subjects With Alzheimer Disease in Comparison to Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Assessment of data shows inadequate brain uptake, suggesting the tracer is inadequate as an imaging biomarker of brain amyloid.
Sponsor: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MNI-168-01
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I 123-MNI-168 (Experimental)
  Interventions: Drug: I-123-MNI-168; Drug: 123-I MNI-168
- I123 MNI168 (Experimental): brain imaging using I123MNI168
  Interventions: Drug: I-123-MNI-168; Drug: 123-I MNI-168

INTERVENTIONS:
Drug: I-123-MNI-168 — Subjects will be injected with up to 5 mCi and not to exceed 5.5 mCi (not >10% of 5 mCi limit) of 123-I MNI-168 followed by serial SPECT imaging.
Drug: 123-I MNI-168 — Subjects will be injected with up to 5 mCi and not to exceed 5.5 mCi (not >10% of 5 mCi limit) of 123-I MNI-168 followed by serial SPECT imaging.

SUMMARY:
The underlying goal of this study is to assess 123-I MNI-168 SPECT imaging as a tool to detect ß-amyloid deposition in the brain of Alzheimer's Disease (AD) research participants and similarly aged and gender matched healthy subjects.

DETAILED DESCRIPTION:
The overall research questions to be addressed by this protocol are as follows:

* To assess the dynamic uptake and washout of (123I) MNI-168, a potential imaging biomarker for β-amyloid burden in brain, using single photon emission computed tomography (SPECT) in Alzheimer's (AD) subjects and similarly aged and gender matched healthy controls.
* To perform blood metabolite characterization of (123I) MNI-168 in healthy and AD subjects to determine the metabolic fate and nature of metabolites in assessment of (123I) MNI-168 as a single photon computed tomography (SPECT) brain imaging agent.
* To acquire initial safety data following injection of (123I) MNI-168.
* Obtain test/retest reproducibility information in AD subjects with (123I) MNI-168 based on initial studies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have a clinical diagnosis of AD will be recruited for this study
* The participant is 50 years or older
* Written informed consent is obtained
* Participants have a clinical diagnosis of probable Alzheimer's disease based on National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria
* Subjects will have a clinical dementia rating (CDR) assessment score of ≥ 0.5 and < 2.0
* Modified Hachinski Ischemia Scale score of ≤ 4
* For females, non-child bearing potential or negative urine and blood pregnancy test on day of 123-I MNI-168 injection

Exclusion Criteria:

* The subject has signs or symptoms of another neurodegenerative disease including Parkinson's disease, diffuse Lewy body dementia, or history of significant cerebrovascular disease
* The subject has clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
* The subject has any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including gastrointestinal surgery)
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease
* The subject has participated in another clinical study within the previous 30 days
* Clinically significant MRI evidence of vascular disease or alternative neurologic disorder
* Pregnancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To assess the uptake and washout of {I123}MNI-168, a potential imaging biomarker for β-amyloid burden in brain, | 1 year

SECONDARY OUTCOMES:
To acquire initial safety data following injection of (123I) MNI-168. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Danna Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States